## Statistical Analysis Cover Page

Study Title: Nicotinamide Riboside in LVAD Recipients (PilotNR-LVAD)

## NCT Number Document Description Document Date

NCT03727646

November 18, 2018

| Statistical Analysis Template ClinicalTrials.gov | | |
|---|---|---|
| Statistical<br>Analysis<br>Overview | * Comparison Group Selection ① | □ Arm/Group 2 □ Arm/Group 3 |
| | Comments ② | We performed a Pre- and Post-NR intervention comparison |
| | * Type of Statistical Test | (Select One) Superiority Equivalence Non-inferiority Qther (for example, single group or other descriptive analysis) |
| | [*] Comments ③ | |
| Statistical Test of Hypothesis | [*] P-Value (if applicable) | 0.0405 (calculated value, not the a priori threshold for statistical significance) |
| | Comments ② | We performed a pairwise 2-tailed student's T-test to compare the Pre-NR and Post-NR PBMC Maximal Respiration |
| | [*] Method<br>(required if p-value entered) | (Select One) ANCOVA Fisher Exact Mixed Models Analysis t-Tes (1-Sided ANOVA Kruskal-Wallis Regression, Cox t-Test, 2-Sided Chi-Squared Log Rank Regression, Linear Wilcoxon Chi-Squared, Corrected Mantel Haenszel Regression, Logistic (Mann-Whitney) Cochran-Mantel-Haenszel McNemar Sign Test Other () |
| | Comments ② | |
| Method of Estimation | [*] Estimation Parameter<br>(if applicable) | (Select One) Cox Proportional Hazard Mean Difference (Net) Odds Ratio, Log Slope Hazard Ratio (HR) Median Difference (Final Values) Risk Difference (RD) Other Hazard Ratio, Log Median Difference (Net) Risk Ratio (RR) () Mean Difference (Final Values) Odds Ratio (OR) Risk Ratio, Log |
| | Estimated Value | (calculated value) |
| | Confidence Interval<br>(if applicable) | Level: % Confidence Interval Number of Sides: (Select One) 2-sided 1-sided Lower Limit: Upper Limit: |
| | Parameter Dispersion | Type: (Select One) Standard Deviation Standard Error of the Mean Value: |

\* Required [\*] Conditionally required

**Other Statistical** Analysis (4)

Estimation Comments (2)

- Use the checkboxes to select the Arms/Groups (pre-populated from the Outcome Measure) involved in the statistical analysis.
- (2) (Optional) Include any relevant information about the row above (e.g., the null hypothesis, details of the power calculation, adjustment for multiple comparisons, the a priori threshold for statistical significance, the direction of the comparison). Do not include written results or conclusions.
- (3) If a non-inferiority or equivalence analysis, information on the definition of the non-inferiority or equivalence margin is required. 4 If the statistical analysis cannot be submitted using the Statistical Test of Hypothesis or Method of Estimation options, provide a description and the results of the scientifically appropriate test of statistical significance.

## Statistical Analysis Plan (SAP)

Given the study is an open label single-arm interventional study without a control group, the change of attributes (whole blood NAD/NR levels, PBMC pro-inflammatory cytokine expression levels, mitochondrial oxygen consumption rate) of each study subject before and after intervention (oral nicotinamide riboside) will be analyzed by the pairwise Student's t-test. If the distribution of the data passes the normality test, a parametric t-test will be used.